CLINICAL TRIAL: NCT01050244
Title: The Effect of Soy Protein on Neuropathic Pain: Randomized N-of-1 Trials
Brief Title: The Effect of Soy Protein on Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ran out_difficulties with study product (delays in authorization).
Sponsor: Dr. Yoram Shir (Other)
Collaborators: Louise & Alan Edwards Foundation (Unknown); McGill University (Other)
Responsible Party: Sponsor-Investigator, Dr. Yoram Shir, Doctor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN 09-117
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Neuralgia
Keywords: Soy protein; Milk protein; Neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy Protein (Experimental): 30g of soy protein from whole soybean soymilk powder given daily for 3 weeks
  Interventions: Dietary Supplement: Whole soybean soymilk powder
- Milk Protein (Placebo Comparator): 30g of milk protein from whole milk powder given daily for 3 weeks
  Interventions: Dietary Supplement: Whole milk powder

INTERVENTIONS:
Dietary Supplement: Whole soybean soymilk powder
  Other Names: Benesoy organic soymilk powder; Code #1386
  Arms: Soy Protein
Dietary Supplement: Whole milk powder
  Other Names: Parmalat Code #202006
  Arms: Milk Protein

SUMMARY:
Neuropathic pain is one form of chronic pain lacking effective pharmacotherapy. Interest in the role of complementary and alternative medicine is growing and diet is at the forefront of the search for alternative treatments for pain. Soy protein is one of the most promising dietary ingredients tested for its pain-relieving properties. Results from animal studies show that soy-enriched diets reduce pain due to nerve injury. The purpose of this study is to determine the effects of soy protein supplementation on facial pain.

DETAILED DESCRIPTION:
Neuropathic pain is a complex disorder with mixed results in response to pain medication due to a high degree of variability between patients. To address this issue, we are implementing a unique methodology using a series of N-of-1 or single subject randomized, double blind, controlled studies. With this, we will explore the role of soy protein supplementation in neuropathic pain patients. Each patient will be exposed in 3-week intervals to soy protein and a control, milk protein, in three paired treatment periods for a total of 18 weeks. This method allows for the measurement of treatment efficacy in individual distinct patients and has the potential for immediate and continued medical benefit using a simple and readily available dietary ingredient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years old
* Chronic neuropathic pain with tactile allodynia > 6 months
* Suboptimal pain pharmacotherapy (i.e. additional pain control felt by patient and physician to be necessary)
* Pain intensity score ≥ 5 on 11-point numerical rating scale (NRS) during 1-week screening period prior to randomization
* Stable medication use (if any) over 4 weeks before starting the trial. Current medication use will be maintained and no additional pharmacotherapy may be introduced during the trial.
* Up to date mammogram and gynecological evaluations.

Exclusion Criteria:

* History of significant heart, gastro-intestinal, liver or kidney disease
* History of alcohol/narcotic abuse or current excessive alcohol consumption
* History or diagnosis of cancer
* History of breast tumors, predisposition to breast cancer or a family member with breast cancer
* History of hormonal or gynaecological disease
* Current use of hormonal replacement therapy (HRT), except thyroid HRT
* Pregnant or breastfeeding women
* Use of any anticoagulant or blood thinner except acetylsalicyclic acid
* Malabsorption of any kind
* Diagnosed lactase deficiency;
* Known allergy to any of the dietary products
* Known allergy to acetaminophen
* Daily consumption of soy protein in quantities exceeding 10 g/day
* Strict vegetarians (i.e. no animal derived dietary sources)
* Antibiotic use within the last 3 months
* Any previous psychiatric diagnosis before pain onset
* Body mass index > 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline and 3 times during the last week of every treatment period

SECONDARY OUTCOMES:
Pain Quality | Baseline and 3 times during the last week of every treatment period
Dynamic tactile allodynia | Baseline and at the end of every treatment period
Area of dynamic allodynia | Baseline and at the end of every treatment period
Quality of life | Baseline and at the end of every treatment period
Depression | Baseline and at the end of every treatment period
Dietary intake | Baseline, once a week during the first treatment period, once during the second week of the remaining treatment periods.
Body weight | Baseline and at the end of every treatment period
Analgesic medication use | Baseline and 3 times during the last week of every treatment period
Adverse events | The full 18 weeks until the end of the last treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Shir, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada